CLINICAL TRIAL: NCT03042897
Title: Endometrial Cancer and Obesity: An Exercise and Diet Intervention for Weight Loss
Brief Title: Exercise and Diet Intervention in Promoting Weight Loss in Obese Patients With Stage I Endometrial Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5U-16-1; NCI-2016-01684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5U-16-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Estrogen Receptor Positive; Obesity; Progesterone Receptor Positive; Stage I Uterine Corpus Cancer; Stage IA Uterine Corpus Cancer; Stage IB Uterine Corpus Cancer
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (exercise and diet) (Experimental): Patients undergo aerobic exercise thrice weekly over 95 minutes for up to 16 weeks. Patients also undergo multi-lifestyle interventions based on the DASH diet once weekly over 1 hour for up to 16 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Undergo DASH diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Behavioral: Exercise Intervention — Undergo in aerobic exercise
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies exercise and diet intervention in promoting weight loss in obese patients with stage I endometrial cancer. Exercise and diet may cause weight loss and minimize the risk of gynecologic surgery related to being overweight in patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if participation in a 16-week exercise and diet intervention would elicit weight loss, assessed by a 10% decrease in fat mass, in endometrial cancer (EC) patients.

SECONDARY OBJECTIVES:

I. To determine if participation in a 16-week exercise and diet intervention would improve cardiorespiratory fitness (CRF) and muscular strength.

TERTIARY OBJECTIVES:

I. To determine if participation in a 16-week exercise and diet intervention could improve quality of life (QOL), fatigue, and depression.

II. To determine the effects of a 16-week exercise and diet intervention on cardiovascular (CV) health.

OUTLINE:

Patients undergo aerobic exercise thrice weekly over 95 minutes for up to 16 weeks. Patients also undergo multi-lifestyle interventions based on the dietary approaches to stop hypertension (DASH) diet once weekly over 1 hour for up to 16 weeks.

After completion of study, patients are followed up for 16 weeks.

After completion of study, patients are followed up for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I EC
* Low grade disease positive for estrogen and progesterone receptors
* Body mass index (BMI) >= 30 kg/m^2
* No history of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise
* Self ambulatory and without use of assistive walking devices
* Is not a candidate for immediate hysterectomy, following evaluation by a physician, due to desire to preserve fertility, due to degree of obesity, due to comorbidities, or due to patient refusal of hysterectomy
* Must agree to take progestin agents (i.e., oral agents or MIRENA intrauterine device [IUD] which are accepted treatments for low grade uterine malignancies to control their disease while the intervention is ongoing)

  * Note: potential participants WILL NOT be asked to delay surgery to participate in this pilot study

Exclusion Criteria:

* Patients with metastatic disease
* BMI =< 29.9 kg/m^2
* History of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise
* Is not self ambulatory and relies on the use of assistive walking devices
* Is a candidate for immediate hysterectomy, following evaluation by a physician
* In judgement of a physician, is not a candidate for progestin agents

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (CRF) | Up to 34 weeks
  Subjects will be instructed to walk comfortably (so they are able to talk while walking) on a treadmill for 4 minutes and heart rate will be measured at the end of the test to estimate maximal oxygen uptake.
Cardiovascular (CV) health outcomes | Up to 34 weeks
  Carotid Intima Media Thickness (cIMT) of the right common carotid artery will be measured using B-mode ultrasound. The ultrasound scan of cIMT provides lumen diameter, intima-media thickness, and presence and extent of plaques.
Depression measured by Center for Epidemiologic Studies Depression scale | Up to 34 weeks
  Will be assessed on a continuum scale and thus our current plan is to use paired t tests. All analysis will be performed using SPSS (v.21).
Fatigue measured by the Brief Fatigue Inventory | Up to 34 weeks
  Will be assessed on a continuum scale and thus our current plan is to use paired t tests. All analysis will be performed using SPSS (v.21).
Muscle strength | Up to 34 weeks
  The 10-repetition maximum (10-RM) method will test maximal voluntary strength for the following exercises: chest press, seated row, knee extension, knee flexion will be used to calculate maximum strength values for the resistance exercise intervention.
Percent weight loss at the completion of the intervention | At 16 weeks
  Each of the 25 women will be classified as having achieve the 10% weight-loss or not. Of those subjects who achieve a weight-loss of 10% or more, the proportion of patients who maintain this weight-loss will also be calculated. The mean percent weight loss, as well as the range and quartiles will be calculated. In addition, for those subjects who fail to achieve a 10% weight-loss, the reasons for failure will be examined (e.g. inability to complete 16 weeks, inability to adhere to the diet, inability to adhere to the exercise schedule, etc.). This information will guide the design (or redesign of the weight loss program as well as the follow-up studies.
Quality of Life (QOL) | Up to 34 weeks
  The SF-36 short-form health survey with 36 items will be used to assess physical and mental health. The FACT-En questionnaire will also be used. This is a 43-item questionnaire including questions regarding the physical well-being, social/family well-being, and additional concerns on the effect of endometrial cancer on the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States